CLINICAL TRIAL: NCT00125775
Title: Phase 4 Study of Recombinant Hepatitis B Vaccine in Peritoneal Dialysis Subjects
Brief Title: Does Extra-High Dose Hepatitis B Vaccination Confer Longer Serological Protection in Peritoneal Dialysis Patients?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr. Kai Ming CHOW, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRE-2005.134
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-07

CONDITIONS: Peritoneal Dialysis; Renal Disease, End-Stage
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Engerix-B 40 mcg dose
  Interventions: Biological: Engerix-B
- 2 (Active Comparator): Engerix-B 80 mcg dose
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: Engerix-B — Engerix-B at 0, 1, 6 months

SUMMARY:
Hepatitis B virus causes inflammation of the liver which is detrimental to the end-stage renal disease patients on dialysis. Hepatitis B vaccine is recommended for this high-risk population although the vaccine protection remains suboptimal and does not last long.

The purpose of this study is to determine the best vaccination strategy over a 6-month period using recombinant hepatitis B vaccine (Engerix-B) in peritoneal dialysis patients. Current data show that the traditional Engerix-B vaccine dose (40 micrograms) does not always lead to protective and long-lasting hepatitis B surface antibody. The investigators, therefore, decided to compare the usual 40-micrograms with an 80-microgram dose strategy of vaccine protection.

DETAILED DESCRIPTION:
The objective of the present randomized study is to evaluate the optimum strategy of recombinant hepatitis B vaccination in the maintenance of protective anti-HBs antibody among end-stage renal disease patients on peritoneal dialysis. This study is designed to establish whether a three-dose schedule of 80 microgram Engerix-B vaccine could maintain protective antibody response among dialysis patients. The secondary aim is to identify the effects of dosing on various subgroups of dialysis patients.

Viral hepatitis B infection remains a major health hazard for end-stage renal disease patients on dialysis. The direct costs of hepatitis B infection and long term impact on morbidity and renal transplantation are substantial. Apart from the devastating consequences of hepatitis B infection on patients on dialysis or after transplantation, infected patients are potential reservoirs for infecting other patients and haemodialysis staff. Antibody production achieved in renal patients is suboptimal; the most effective method of vaccination to prevent hepatitis B infections in end-stage renal disease subjects has hitherto been unanswered by the current literature and the latest Cochrane Collaboration review.

Given the relatively low seroconversion rate and maintenance of protective hepatitis antibody levels among end-stage renal disease patients, a treatment strategy using various doses of recombinant hepatitis B vaccine (Engerix-B) has been recently explored. In an observational study, the investigators demonstrated no statistically significant difference in response rate between patients receiving three recommended doses of Engerix-B intramuscularly (40 micrograms each dose) and those with four times the normal adult dose (80 micrograms each dose), (78% versus 100%, P = 0.23). On the other hand, according to the Kaplan-Meier estimates, 78 percent of patients in the 40 micrograms Engerix-B vaccination group and 96 percent of patients in the 80 micrograms dosing group had maintained the seroprotective levels of antibody to hepatitis B surface antigen (anti-HBs) at 12 months after initial response. This difference corresponds to an absolute risk reduction of 18 percent for losing the antibody response with a three-dose schedule of 80 micrograms Engerix-B vaccination program. In other words, the investigators estimate that giving Engerix-B 80 micrograms dose would lead to one extra end-stage renal disease subject with persistent seroprotective anti-HBs level at one year for every 5.6 patients treated (number needed to treat to benefit NNT, 5.6; 95% confidence interval, 5.4 to 5.8).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* End-stage renal disease and on maintenance peritoneal dialysis
* Serologically negative for hepatitis B surface antigen (HBsAg) and antibody to hepatitis core antigen (anti-HBc)
* No history of receiving hepatitis B vaccination
* Willingness to give written informed consent and willingness to participate in and comply with the study protocol

Exclusion Criteria:

* Expected survival less than 6 months
* Those who refused vaccination
* Active malignancy
* Alcoholic liver disease
* Chronic hepatitis C and/or human immunodeficiency virus (HIV) infection
* Receiving immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
hepatitis B surface antibody anti-HBs level ≥ 10 IU/L 3 months after completion of the third dose and the persistence of protective anti-HBs 12 months after completion of the third dose of Engerix-B vaccine | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Chow, MRCP, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, New Territories, New Territories, Hong Kong